CLINICAL TRIAL: NCT02778009
Title: Fit Physicians: A Novel Physical Activity Integration Program to Improve Fitness and Activity in Medical Students: A Randomized Pilot Study
Brief Title: Fit Physicians: Use of Activity Monitors and Activity Integration Program in First Year Medical Students
Acronym: FitPhysician
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Joanne DiFrancisco-Donoghue, Assistant Professor, Ph. D., New York Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BHS-1153
Record Dates: First submitted 2016-04-08; First posted 2016-05-19 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Motor Activity; Body Weight Changes
Keywords: Medical student; Activity Monitor; Medical school; Fitness
MeSH Terms: conditions — Motor Activity; Body Weight Changes | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fit Physician Group (Experimental): Subjects will receive activity monitor and will be required to attend monthly wellness lectures and weekly exercise intervention.
  Every subject will undergo an iDEXA scan to measure body mass composition
  Interventions: Radiation: iDEXA Scan; Other: Wellness Lectures; Other: Exercise intervention; Other: Activity monitor
- Activity Monitor Only Group (Active Comparator): Subjects will receive an activity monitor without any intervention Every subject will undergo an iDEXA scan to measure body mass composition
  )
  Interventions: Radiation: iDEXA Scan; Other: Activity monitor
- Control Group (Other): Subjects will not an activity monitor nor will they receive any intervention Every subject will undergo an iDEXA scan to measure body mass composition
  Interventions: Radiation: iDEXA Scan

INTERVENTIONS:
Radiation: iDEXA Scan — Subjects will receive pre study and post study scans to assess body mass composition
Other: Wellness Lectures — Subjects in the Fit Physician Arm will be required to attend monthly wellness lectures
  Arms: Fit Physician Group
Other: Exercise intervention — Subjects in the Fit Physician Arm will be required to attend weekly exercise interventions
  Arms: Fit Physician Group
Other: Activity monitor — Subjects in the Fit physician arm and the activity monitor arm will receive activity monitors to assess their activity level throughout the academic year
  Arms: Activity Monitor Only Group; Fit Physician Group

SUMMARY:
Using FitBit activity monitors, physical activity levels will be monitored in first year medical students. Body Composition will be measured as well.

DETAILED DESCRIPTION:
Using fitness trackers and exercise testing, it will determine if participating in a novel program that incorporates wellness into the academic term will improve fitness.

An estimate, 120 students will enroll in this study. Men and women aged 18-55 years of age that are just entering medical school. Students who are currently pregnant will not be allowed to participate in this study.

Participation will involve 2 visits at the start of the academic school year, and two visits at the end of the academic school year.

These visits will entail you undergoing a body composition scan measured by an duel energy x-ray absorptiometry (iDEXA) machine. The scan takes approximately 15 minutes. Subjects may be asked to perform an exercise stress test on a treadmill. The exercise test is approximately 40 minutes. Subjects may be asked to participate in a fitness program 2x a week, and may be asked to wear a Fitbit Flex™ activity tracker on the wrist for the duration of the school year. Investigators will be accessing academic grades to use for statistical purposes only. Subject names will never be given to any other party other than the investigators involved.

ELIGIBILITY:
Inclusion Criteria:

* First year medical students
* Must have smartphone

Exclusion Criteria:

* Medical conditions that prohibit exercise
* pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2017-06-03 (Actual); Study Completion 2017-06-03 (Actual)

PRIMARY OUTCOMES:
Steps per day measured daily by FitBit Flex | 10 months

SECONDARY OUTCOMES:
Body Mass Composition assessed by iDEXA scan | 10 months
Academic Performance assessed by numeric grade point average | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian Harper, MD, Study Chair — NYIT College of Osteopathic Medicine
Locations (1):
- NYIT, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with individual participants

REFERENCES:
- [Derived] DiFrancisco-Donoghue J, Jung MK, Stangle A, Werner WG, Zwibel H, Happel P, Balentine J. Utilizing wearable technology to increase physical activity in future physicians: A randomized trial. Prev Med Rep. 2018 Sep 11;12:122-127. doi: 10.1016/j.pmedr.2018.09.004. eCollection 2018 Dec. PMID 30234000